CLINICAL TRIAL: NCT07001735
Title: Talking for Change: A Patient Preference Randomized Controlled Trial
Brief Title: Talking for Change: Secondary Prevention of Child Sexual Abuse Perpetration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Cory Gerritsen, Collaborating Scientist, Slaight Centre for Early Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/178
Record Dates: First submitted 2025-03-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Pedophilia; Hebephilia; Child Sexual Abuse; Program Evaluation; Prevention Intervention; Paraphilias and Paraphilic Disorders
Keywords: paraphilias; group psychotherapy; child sexual abuse; sexual offending against children; prevention; crime prevention; psychotherapy; dynamic risk factors; pedophilia; hebephilia; mechanisms of change; protective factors; individuals with sexual interest in children; forensic psychology; preventive psychiatry; Internet based intervention
MeSH Terms: conditions — Pedophilia; Paraphilic Disorders

STUDY DESIGN:
Intervention Model Description: Three-armed preference trial with active psychological placebo control and non-randomized no-intervention control arm; placebo control participants will receive experimental treatment after placebo and vice-versa
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Natural History Benchmarking (No Intervention): A subset of participants will participate in a video-conferencing interview and will complete an online survey comprising self-report measures at two time points, 20 weeks apart.
  A subset of participants will complete an online survey comprising self-report measures at two time points, 20 weeks apart.
- General Mental Health Group Psychotherapy (Active Comparator): The active therapeutic control is a general mental health intervention that is not specific to managing risk for child sexual abuse perpetration.
  Interventions: Behavioral: Healthier Me: Managing Risk and Stress in Everyday Life
- Talking for Change (TFC) Group Psychotherapy (Experimental): Talking for Change (TFC) is a secondary prevention program that targets dynamic risk factors for child sexual abuse perpetration.
  Interventions: Behavioral: Talking for Change Group Psychotherapy

INTERVENTIONS:
Behavioral: Talking for Change Group Psychotherapy — Talking for Change (TFC) is a secondary prevention program that targets dynamic risk factors for child sexual abuse, including (1) atypical sexual interests and sexual self-regulation problems; (2) problems in relationships; (3) offense-supportive attitudes; and (4) general self-regulation deficits and related traits (e.g., impulsivity, emotion regulation deficits). Participants will complete 20 weekly, 120-minute sessions delivered via WebEx.
  Arms: Talking for Change (TFC) Group Psychotherapy
Behavioral: Healthier Me: Managing Risk and Stress in Everyday Life — The active therapeutic control is a non-directive supportive psychotherapy that targets general mental health concerns. It consists of psychoeducation about human sexuality and common mental health concerns, as well as instruction and practice in applied relaxation and stress management, and group discussions that will facilitate sharing and problem-solving current stressors. This active control intervention is equivalent in length to Talking for Change (TFC), consisting of 120-minute long occurring weekly over the course of 20 weeks.
  Arms: General Mental Health Group Psychotherapy

SUMMARY:
The goal of this patient preference randomized controlled trial is to investigate the efficacy of Talking for Change (TFC), an intervention for the secondary prevention of child sexual abuse and exploitation (CSA) perpetration. Blinded clinical raters will evaluate the primary endpoint-reductions in dynamic risk factors for sexual offending against children-and clients will provide self-reports to evaluate a second primary outcome-reductions in sexual contact with children, accessing online child sexual exploitation material (CSEM), and desire for sexual contact with children. Researchers will compare the following groups: (1) those receiving 20 weeks of the experimental TFC group psychotherapy; (2) those receiving 20 weeks of a control group psychotherapy targeting mental health and stress more broadly; and (3) those receiving no treatment.

DETAILED DESCRIPTION:
Child sexual abuse (CSA) is a preventable public health issue that has significant mental health, physical health, financial, societal, and personal consequences. In Canada, perpetration prevention interventions are typically provided after CSA has occurred and its damaging sequelae have already occurred (i.e., tertiary prevention interventions are provided to those already convicted to prevent re-offending). These tertiary prevention interventions are reactive in nature and represent one form of the prevention spectrum.

One approach to CSA perpetration prevention that has been historically neglected in Canada is secondary prevention. Secondary CSA perpetration prevention interventions aim to prevent the onset of CSA perpetration by targeting populations that are at elevated risk. These interventions focus on helping at-risk adults understand and manage psychosocial risk factors that are causes of CSA perpetration. By targeting these risk factors, secondary perpetration prevention treatment programs help at-risk individuals live offense-free lives. At present, there is a lack of data on whether secondary CSA perpetration prevention programs are efficacious in reducing CSA perpetration.

Talking for Change (TFC) is a secondary CSA perpetration prevention intervention offering psychotherapy to adults who are concerned about their risk of perpetrating CSA or accessing online child sexual exploitation material (CSEM). The target client population of TFC are adults with a sexual interest in children, those who self-identify as being at-risk of viewing CSEM, or those who self-identify as at-risk of having sexual contact with children. TFC targets dynamic risk factors that are the causes of engaging in CSA or accessing CSEM, including (1) atypical sexual interests and sexual self-regulation problems; (2) problems in relationships; (3) offense-supportive attitudes; and (4) general self-regulation deficits and related traits (e.g., impulsivity, emotion regulation deficits).

The primary objective of the proposed research is to examine the efficacy of TFC via a patient preference randomized controlled trial to test superiority over (a) active psychological control and (b) no-treatment control arms. More specifically, the present trial aims to understand whether TFC produces significantly greater improvement in established risk factors for CSA perpetration and reductions in CSA behavior compared to the two control arms.

The secondary objectives of the research are to examine additional outcomes (including quality of life and treatment indicators) and examine mediators of treatment change. These secondary outcomes will allow for a more fulsome understanding of the effects of TFC and insight into mechanisms of change in TFC.

This is a single-blind patient preference randomized controlled trial of TFC versus active control, with a third non-randomly allocated no treatment control arm (i.e., a natural history benchmarking arm). Briefly, eligible clients referred to TFC who consent to participate in the trial will first be asked if they are willing to be randomized into one of the two trial treatment arms. Those who decline to be randomized will enter the study arm they prefer. The advantage of this approach is that it can accommodate the methodological rigor associated with a randomized clinical trial while reducing trial non-participation among those with a strong treatment preference. Once clients complete one arm of the trial, they will be offered the opportunity to participate in the second arm of the trial. In either case, continuation into the alternate intervention will be optional as will the continued collection of study data.

Benchmarking for natural history processes will involve data collection on online forums for individuals with pedohebephilic interests (i.e., those with an attraction to prepubescent and pubescent minors). Participants in the benchmarking arm will be involved in two assessment time points over the course of 20 weeks, which will allow for estimating change on primary and secondary outcomes over a period of time equivalent to the duration of the TFC and control treatment arms of the trial. Inclusion of a benchmarking sample allows the researchers to compare the effect of TFC to natural history processes (e.g., maturation, the passage of time).

Two groups of benchmarking participants will be recruited, with participants in the two groups receiving a different assessment battery. The first group will complete an online survey of self-report measures and a psychosocial interview focused on risk factors for sexual offending and protective factors. Once an adequate number of benchmarking participants have completed an interview, recruited participants will complete only the online survey containing self-report measures. The decision to use this stopping rule for the benchmarking arm was based on power analyses using effect size data from a pilot evaluation of the TFC program.

ELIGIBILITY:
INCLUSION CRITERIA:

For the treatment arms, the participant must meet all of the inclusion criteria to eligible for this clinical trial:

1. Must be deemed to have capacity to provide informed consent;
2. Must sign and date the informed consent form;
3. Stated willingness to comply with all study procedures;
4. Be 18 years of age or older upon study commencement;
5. Be referred for care in the TFC program due to concerns about enhanced risk of sexual offending against children.

For the benchmarking interview arm, the participant must meet all of the following inclusion criteria:

1. Must self-report concerns about enhanced risk of sexual offending against children
2. Must be deemed to have capacity to provide informed consent;
3. Must check the appropriate box on the informed consent form;
4. Stated willingness to comply with all study procedures;
5. Be 18 years of age or older upon study commencement.

For the benchmarking survey arm, participants must check the appropriate box on the informed consent form.

EXCLUSION CRITERIA:

For the treatment arms:

1. Inability to engage meaningfully in group psychotherapy (e.g., due to intellectual disability, other neurodiversity, active psychosis or substance use)
2. Those who self-identify as at-risk for reasons better accounted for by non-risk-relevant factors per clinical assessment (e.g., those with obsessive-compulsive disorder including thoughts about CSA, who commonly fear that they are at-risk but are not).
3. Non-male sex.

For the benchmarking interview arm:

1. Non-male sex.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The sample for this study will consist of individuals who were assigned male at birth.
Enrollment: 220 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Violence Risk Scale - Sexual Offense Version (VRS-SO) | Treatment arm: pre-treatment (within 4 weeks of starting) and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  24 items (7 static and 17 dynamic risk factors) rated on a scale from 0 to 3; higher scores indicate higher risk; total static scores range from 0 to 21; total dynamic scores range from 0 to 51; dynamic risk factors rated 2 or 3 are designated treatment targets; each treatment target is further rated in terms of readiness for change (pre-contemplation, contemplation, preparation, action, and maintenance).

SECONDARY OUTCOMES:
Structured Assessment of Protective Factors against Sexual Offending (SAPROF-SO) | Treatment arm: pre-treatment (within 4 weeks of starting) and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  14 items (and 6 additional optional items) rated on a scale from 0 to 4; higher scores indicate greater presence of the protective factor; total scores range from 0 to 56 (80, if the optional items are included).
Frequency of Use of Illegal Child Sexual Abuse Imagery | Treatment arm: Pre-treatment (within 4 weeks of starting) and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  4 items rated on a 5-point Likert scale; higher scores indicate more frequent consumption of sexual imagery of children; total scores range from 4 to 20.
Frequency of Desire for Sexual Activities with Minors | Treatment arm: Pre-treatment (within 4 weeks of starting) and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  4 items rated on a 5-point Likert scale; higher scores indicate greater desire to engage in sexual contact with minors; total scores range from 4 to 20.
Frequency of Sexual Activities with Minors | Treatment arm: Pre-treatment (within 4 weeks of starting) and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  3 items on a 5-point Likert scale; higher scores indicate greater frequency of one's sexual contact with minors; total scores range from 3 to 15.
Coping Using Sex Inventory (CUSI) | Treatment arm: pre-treatment (within 4 weeks of starting), Treatment Week 10, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  8 CUSI items, rated on a 5-point Likert scale, will be used in this trial; higher scores indicate greater tendency to use sex to cope with problematic situations; total scores range from 8 to 40.
Compulsive Sexual Behavior Inventory - 13 (CSBI) | Pre-treatment (within 4 weeks of starting), Treatment Week 10, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  13 items rated on a 5-point Likert scale; higher scores indicate greater sexual compulsivity; total scores range from 13 to 65.
Cognitions that Support Sexual Offending Against Children Scale - Short Form (CSSOC-SF) | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 10, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  10 items rated on a 4-point Likert scale; higher scores indicate greater endorsement of cognitions that support and condone sexual offending; total scores range from 10 to 40.
Children and Sex Questionnaire: Emotional Congruence with Children | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 10, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Week 1 and Week 20.
  3 items from this scale, rated on a 4-point Likert scale, will be used in this trial; higher scores reflect greater emotional congruence with children; total scores range from 3 to 12.
Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 10, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  18 items rated on a 5-point Likert scale; higher scores indicate greater difficulties with emotion regulation; total scores range from 18 to 90.
Aggression Inventory (AI) | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 10, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  9 items rated on a 5-point Likert scale; higher scores indicate greater aggression; total scores range from 9 to 45.
Brief Aggression Questionnaire (BAQ) | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 10, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  6 items from this measure, rated on a 7-point Likert scale, will be used in this trial; higher scores indicate greater aggression; total scores range from 6 to 42.
Problems in Interpersonal Relationships | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 10, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  22 items rated on a 4- to 7-point Likert scale; higher scores indicate greater loneliness, social isolation, and experience of jealousy in intimate relationships; total scores range from 22 to 134.
Dimensions of Skillfulness and Use Scale (DSUS) | Weekly over the course of the 20 treatment weeks. Repeated for the second treatment.
  4 items rated on a 5-point Likert scale; higher scores indicate greater understanding and use of skills learned in the session; total scores range from 4 to 20.
Clinical Outcomes in Routine Evaluation -10 (CORE-10) | Weekly over the course of the 20 treatment weeks. Repeated for the second treatment.
  10 items rated on a 5-point Likert scale; higher scores indicate more problems with psychological symptoms, functional impairment, and risk to self; total scores range from 0 to 40.
The Multitheoretical List of Therapeutic Interventions 30 | Weekly over the course of the 20 treatment weeks. Repeated for the second treatment.
  30 items rated on a 5-point Likert scale; higher scores indicate higher quality and intensity of interventions provided during therapy sessions; total scores range from 30 to 150.
Curative Climate Instrument (CCI) | Treatment Weeks 1, 7, 14 and 20. Repeated for the second treatment.
  9 items rated on a 4-point Likert scale; higher scores indicate greater presence of therapeutic factors; total scores range from 9 to 36.
Group Climate Questionnaire - Short Form (GCQ-S) | Treatment Weeks 1, 7, 14 and 20. Repeated for the second treatment.
  12 items rated on a 7-point Likert scale; higher scores indicate a more favorable perception of the group therapeutic environment; total scores range from 0 to 72.
Treatment Motivation Questionnaire - Revised (TMQ-R) | Pre-treatment (within four weeks of starting) and at Treatment Week 3. Repeated for the second treatment.
  19 items rated on a 7-point Likert scale; higher scores indicate greater motivation to participate in treatment; total scores range from 19 to 133.
Group Questionnaire - 12 | Treatment Weeks 1, 7, 14 and 20. Repeated for the second treatment.
  4 items from this scale, rated on a 7-point Likert scale, will be used in this trial; higher scores indicate a more positive experience in the therapy group; total scores range from 0 to 24.
Trust and Respect for Clinician Scale (TRCS) | Treatment Weeks 1 and 7. Repeated for the second treatment.
  8 items from this scale, rated on a 7-point Likert scale, will be used in this trial; higher scores indicate greater level of trust and respect for the clinician; total scores range from 8 to 56.
Therapeutic Factors Inventory - Short Form | Treatment Weeks 1, 7, 14 and 20. Repeated for the second treatment.
  13 items from this scale, rated on a 7-point Likert scale, will be used in this trial; higher scores indicate stronger perceptions of four therapeutic factors (instillation of hope, secure emotional expression, awareness of relational impact, and social learning); total scores range from 13 to 91.
Therapeutic Agency Inventory (TAI) | Treatment Weeks 1, 7, 14 and 20. Repeated for the second treatment.
  10 TAI items, rated on a 5-point Likert scale, will be used in this trial; higher scores indicate more experience of agency in therapy; total scores range from 10 to 50.
Relationship Questionnaire (RQ) | Treatment arms: pre-treatment (within 4 weeks of starting). Repeated for the second treatment. Benchmarking arm: Week 1.
  4 items rated on a 7-point scale; higher scores on each item indicate greater identification with the attachment style the item describes; scores for each attachment style range from 1 to 7.
Forms of Self-Criticizing & Self-Reassuring Scale - Short Form (FSCRS-SF) | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 7, Treatment Week 14, post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  14 items rated on a 5-point Likert scale; higher scores indicate a greater sense of inadequacy (scores range from 0 to 20), self-hate (scores range from 0 to 16), and self-reassurance (score scores range from 0 to 20).
Multidimensional Psychological Flexibility Inventory (MPFI) | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 7, Treatment Week 14, post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  45 items from this scale, rated on a 6-point Likert scale, will be used in this trial; higher scores reflect greater psychological flexibility; total scores range from 45 to 270.
Coping Strategy Indicator Short Form (CSI-SF) | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 7, Treatment Week 14, post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  18 items rated on a 3-point Likert scale; higher scores reflect a greater tendency to cope using problem-solving, seeking social support, or avoidance; total scores range from 18 to 54.
CBT Suitability Scale (CBT-SUITS) | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 7, Treatment Week 14, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  13 items rated on a 5-point Likert scale; higher scores indicate greater beliefs and attitudes consistent with cognitive behavioral therapy; total scores range from 13 to 65.
Cognitive and Behavioral Response to Stress Scale | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 7, Treatment Week 14, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  6 items from this scale, rated on a 7-point Likert scale, will be used in this trial; higher scores indicate more frequent cognitive and behavioral responses to stressful or upsetting situations; total scores range from 0 to 36.
General Self-Efficacy Scale | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 7, Treatment Week 14, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  10 items rated on a 4-point Likert scale; higher scores indicate greater self-efficacy; scores range from 10 to 40.
Experience, Understanding, and Management of Risk-Relevant Sexuality | Treatment arms: pre-treatment (within 4 weeks of starting), Treatment Week 7, Treatment Week 14, and post-treatment (within 4 weeks of completing). Repeated for the second treatment. Benchmarking arm: Weeks 1 and 20.
  12 items rated on a 7-point Likert scale; higher scores reflect greater ability to manage one's sexual arousal and behavior in one's daily life; total scores range from 12 to 84.

CONTACTS AND LOCATIONS:
Overall Officials: Artemis Igoumenou, M.D., Ph.D., Principal Investigator — Complex Care and Recovery Program, Centre for Addiction and Mental Health (CAMH); Ian McPhail, Ph.D., C. Psych., Principal Investigator — Bloomberg School of Public Health, Johns Hopkins University; Cory Gerritsen, Ph.D., C. Psych, Principal Investigator — Slaight Centre for Early Intervention, Centre for Addiction and Mental Health (CAMH)
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant survey data will be preserved and made available via controlled access. The data shared will not contain personally identifying information. Data dictionaries will be made available via open access in Open Science Framework (OSF) and the Johns Hopkins Research Data Repository. Controlled access is being proposed to balance protecting participant data, given the sensitivity of the data collected in the study, and facilitating other researchers' access to the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For data shared through a data access agreement, beginning 3 months and ending 5 years following each article publication.
Access Criteria: Sharing access criteria: Investigators who provide a methodologically sound proposal, and whose proposed use of the data has been approved by an independent review committee (e.g., a university ethics review board) identified for this purpose will be provided access.
  Types of analyses: Meta-analytic reviews, analyses that facilitate understanding of the client population and psychotherapeutic processes with these clients.
  How to access IPD: Proposals will be sent to ian.mcphail@jhu.edu, Artemis.Igoumenou@camh.ca, and elizabeth.letourneau@jhu.edu. To be granted access to the data, data requesters will need to sign a data access agreement. Data will be made available digitally via a secure data transfer facility provided by the Centre for Addiction and Mental Health.